CLINICAL TRIAL: NCT02360969
Title: Effect of Neuromuscular Blockade on the Oculomotor by Not Squinting Child
Acronym: STRABO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0908125; 2010-021022-35 (EudraCT Number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Strabismus
Keywords: strabismus; surgical procedure; anesthesia; squint; child
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy subjects waiting for surgery: patients for whom surgery under general anesthesia with administration of curare is planned will be offered an examination of the eyes before and during surgery
  Interventions: Other: Examination of the eye

INTERVENTIONS:
Other: Examination of the eye — Before planed surgery, an ophthalmologist measures the patient's visual acuity and realise an oculomotor examination. Measurement the refraction and the axial length of the eye is performed. Photographs wakefulness are performed.
  During surgery, participation in this study does not involve any change in the course of anesthesia and surgery.
  Pictures of the eye will be performed under general anesthesia.
  Timing photos will be dictated by the values of BIS and train-of-four (TOF). Photos will be conducted at different times, with the "top" given by the anesthetist under the following conditions:
  Deep anesthesia: BIS <50 Deep anesthesia and muscle relaxation: BIS <50 and TOF 0/4

SUMMARY:
Strabismus is a common condition (4-6% of the population) . The screening and treatment is a public health issue. Indeed, beyond the disfigurement, this disease is very supplier of amblyopia which is definitive if it is not detected and treated early (before 6 years old).

Initial treatment of strabismus is medical with orthoptic reeducation through penalization of the better eye in case of amblyopia or wearing optical correction in case of associated refractive disorder.

The second step is the treatment of strabismus is the surgery, when medical treatment has not resulted in a recovery of the visual axes. The principle of surgery is to weaken or strengthen one or more extraocular muscles of one (or two) eye to correct the eyes squint deviation. The main difficulty of surgical treatment is to assess the amount of strengthening or weakening muscles to do in order to obtain the best result and for a long time.

The investigators know that the postmortem anatomical position of the eyes is generally a slight elevation and divergence, but is inferior to the angle of divergence of the orbital axes. Curare and similar products which inhibit the nervous transmission at the neuromuscular junction, can be used to reproduce this situation in normal subjects.

The sign of general anesthesia is then to evaluate the angle of strabismus when the patient is under deep general anesthesia and with a complete muscle relaxation, obtained only when curarised it. If one or both eyes are recovering under general anesthesia, strabismus is mainly due to dynamic changes and surgery limiting muscle play (wire operation) and sometimes one eye is justified. A combination of both is possible (down + wireless), guided by the importance of the sign of general anesthesia on two prominent eyes or one eye. This sign of general anesthesia is however less known and most poorly quantified in healthy subjects. Yet it seems very important to determine what is deviation in normal subjects after neuromuscular blockade, as his eye movement is also subject to mechanical factors and spastic. This would indicate whether the state of rectitude (no strabismus) is the result of a deviation at complete rest (appearing under general anesthesia) and corrected by spastic elements wakefulness or, in another case this righteousness is already present in the state of general anesthesia (due to static factors) and slightly modified by enlightenment.

ELIGIBILITY:
Inclusion Criteria:

* normal visual acuity for age: 10/10 (Test of Cadet) Rossano 2 for 4-6 years old. 10/10 (scale Monoyer) Parnaud 1.5 for 7-15 years old.
* normal oculomotor examination: Examination under normal alternating display eliminating strabismus
* Binocular vision less than or equal to 60 sec/arc for the stereoscopic vision test
* Refraction WITHOUT cycloplegia within normal limits: below 2 dioptries myopia, hyperopia less than 1.5d, below 1 dioptry astigmatism, anisometropia less than 1 dioptry.
* Examination of the fundus without normal pupillary dilation
* Axial length 6 normal for age as measured by noncontact biometer to eliminate refractive offset anomaly axial length by abnormal

Exclusion Criteria:

* presence of anterior eye history
* children whose behavior suggests a poor cooperation when taking photo awakeness
* children with abnormal limb
* scheduled surgery without the use of curare

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients for whom surgery under general anesthesia with administration of curare is planned
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Horizontal deflection of the two eyes under deep general anesthesia and under curare | From the anesthesia to the end of the surgery
  When the patient is under deep general anesthesia (Bispectral Index (BIS) < 50) ,one photo is taken. A seconde one is taken after curare induction.

SECONDARY OUTCOMES:
Horizontal deflection of the two eyes under deep general anesthesia | From the anesthesia to the end of the surgery
  Before the anesthesic induction, one photo is taken. A seconde one is taken when the patient is under deep general anesthesia (Bispectral Index (BIS) < 50)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PM MANOLI, M.D, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No